CLINICAL TRIAL: NCT06908499
Title: Ten-Year Outcomes of Randomized Comparison of Drug-eluting Stent Implantation Versus Optimal Medical Treatment in Patient With Chronic Total Occlusion: DECISION-CTO Trial
Brief Title: The DECISION-CTO Extended 10 Y Follow-up
Acronym: DecisionCTO10Y
Status: Not yet recruiting | Type: Observational
Sponsor: Seung-Jung Park (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, Principal Investigator, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV2025-01
Record Dates: First submitted 2025-04-01; First posted 2025-04-03 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease
Keywords: Chronic Total Occlusion; Drug-eluting Stent Implantation; Optimal Medical Treatment
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with chronic total occlusion: Patients with chronic total occlusion who were enrolled in the original DECISION-CTO trial (NCT01078051)

SUMMARY:
The goal of this clinical trial is to compare long term efficacy of drug-eluting stent implantation compare to optimal medical treatment in patient with chronic total occlusion in a very long-term follow-up (minimum 10 years) period.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical 1) Patients with angina or silent ischemia and documented ischemia 2) Patients who are eligible for intracoronary stenting 3) Age >18 years
2. Angiographic 1) De novo lesion Chronic Total Occlusion (CTO) 2) Reference vessel size ≥ 2.5 mm by visual estimation 3) At least one CTO lesions located in proximal or mid epicardial coronary artery.

   (If the patient has two CTO lesions, one CTO lesion should be located in proximal or mid epicardial coronary artery)
3. CTO definition: TIMI (Thrombolysis in Myocardial Infarction) flow 0 or 1 with estimated duration over 3 months

   * The duration of the occlusion was determined by the interval from the last episode of acute coronary syndrome, or
   * In patients without a history of acute coronary syndrome, from the first episode of effort angina consistent with the location of the occlusion

     1. Angiographically defined total occlusion over 3 months
     2. If no definite symptom with total occlusion, two experienced operators decide CTO in consideration of angiographical morphology (degree of calcification, bridging collaterals, non-tapered stump, angiographic filling from collaterals)

Exclusion Criteria:

1. History of bleeding diathesis or coagulopathy
2. Pregnant state
3. Three vessel CTOs
4. Known hypersensitivity or contra-indication to contrast agent and heparin
5. ST-elevation acute myocardial infarction requiring primary stenting
6. Culprit total occlusion presented with acute coronary syndrome suggesting acute or recent occlusion
7. Characteristics of lesion 1) Left main disease 2) In-stent restenosis 3) Graft vessels 4) Distal epicardial coronary artery CTO lesions 5) Two vessel proximal segment CTOs
8. Hematological disease (Neutropenia <3000/mm3, Thrombocytopenia <100,000/mm3)
9. Hepatic dysfunction, liver enzyme (ALT and AST) elevation ≥ 3 times normal
10. Renal dysfunction, creatinine ≥ 2.0mg/dL
11. Contraindication to aspirin, clopidogrel or other commercial antiplatelet agent
12. Left ventricular ejection fraction <30%
13. Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period.
14. Non-cardiac co-morbid conditions are present with limited life expectancy or that may result in protocol non-compliance (per site investigator's medical judgment).

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with chronic total occlusion who were enrolled in the original DECISION-CTO trial (NCT01078051)
Sampling Method: Non-Probability Sample
Enrollment: 840 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Event rate of the composite event | 10 years
  The composite of all cause death, myocardial infarction, stroke and any revascularization at minimum of 10 years follow-up.

SECONDARY OUTCOMES:
Event rate of all cause death | 10 years
Event rate of myocardial infarction | 10 years
Event rate of stroke | 10 years
Event rate of any revascularization | 10 years

CONTACTS AND LOCATIONS:
Locations (19):
- Ruby Hall Clinic, Pune, Maharashtra, India
- Medistra Hospital, Jakarta, DKI Jakarta, Indonesia
- South Korea (15):
  - SAM hospital, Anyang
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si
  - Dong-A Medical Center, Busan
  - Kangwon National University Hospital, Chuncheon
  - Keimyung University Dongsan Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - The Catholic University of Korea, Daejeon St. Mary's Hosptial, Daejeon
  - Gangneung Asan Hospital, Gangneung
  - Chonnam National University Hospital, Gwangju
  - Bundang CHA Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Hallym University Hangang Sacred Heart Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Ulsan University Hospital, Ulsan
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taipei City, Taiwan
- King Chulalongkorn Memorial Hospital, Bangkok, Thailand